CLINICAL TRIAL: NCT01268722
Title: Balloon Angioplasty Versus Self-expanding Stent for Recanalization of Chronic Total Occlusions of the Femoral Artery
Brief Title: Balloon Angioplasty Versus Primary Stenting for the Treatment of Femoropopliteal Artery Chronic Total Occlusions
Acronym: FACTORY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, SIABLIS DIMITRIOS, Professor of Radiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30357/2-12-2010
Record Dates: First submitted 2010-12-02; First posted 2010-12-31 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Total Occlusion of Artery of the Extremities
Keywords: Nitinol Stent; Balloon angioplasty; Chronic total occlusions; Femoropopliteal
MeSH Terms: interventions — Angioplasty, Balloon; Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balloon (Active Comparator)
  Interventions: Device: Balloon angioplasty
- Stent (Experimental)
  Interventions: Device: Primary stenting

INTERVENTIONS:
Device: Balloon angioplasty — This arm will include patients randomized to undergo the treatment of a chronic total occlusion of the femoropopliteal artery with the use of balloon angioplasty
  Other Names: Percutaneous angioplasty; Balloon dilatation
  Arms: Balloon
Device: Primary stenting — This arm will include patients randomized to undergo primary stenting of the femoropopliteal chronic total occlusion
  Other Names: Self-expandable; Nitinol stents
  Arms: Stent

SUMMARY:
This is a multicenter double-arm randomized trial investigating plain balloon angioplasty versus primary placement of self-expanding nitinol stents after endovascular recanalization of femoral CTOs. Study will recruit up to 200 patients to be adequately powered for detection of a significant difference in vessel patency after 1 year.

DETAILED DESCRIPTION:
Primary placement of new-generation nitinol stents compared to plain old balloon angioplasty has shown encouraging long-term results in the femoropopliteal artery. However, there is complete lack of data about performance of new-generation nitinol stents in the treatment of chronic total occlusions (CTO) of the Femoral artery. This is a multicenter double-arm randomized trial investigating plain balloon angioplasty versus primary placement of self-expanding nitinol stents after endovascular recanalization of femoral CTOs. Study will recruit up to 200 patients to be adequately powered for detection of a significant difference in vessel patency after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 30 years, both genders, no healthy volunteers
* Negative pregnancy test for women of childbearing age
* Symptomatic leg ischemia by Rutherford/Becker Classification (category 3, 4 or 5), i.e. lifestyle-limiting claudication or critical limb ischemia Single completely occluded de-novo superficial femoral artery lesion (femoral artery CTO target lesion)
* Combined overall length of treatable occluded SFA lesion >/= 4.0 cm to </= 15.0 cm, by visual estimate. The occlusion must be treatable with no more than two stents, minimizing the stent overlap.
* Randomization process before successful subintimal or intraluminal recanalization of the lesion in order to evaluate technical success
* Use of re-entry devices at the discretion of the operator
* All lesions are to be located at least three centimeters (3 cm) proximal to the superior edge of the patella
* Reference vessel diameter (RVD) >/= 4.0 mm and </ 6.0 mm by visual assessment
* At least 1 patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (< 50% stenosis) to the ankle or foot
* Poor aortoiliac or common femoral "inflow" (i.e. angiographically defined > 50% stenosis of the iliac or common femoral artery) lesions must be successfully treated prior to treatment of the target lesion
* Bilateral obstructive SFA disease is eligible for enrollment into the study
* Patient or authorized representative must provide written informed consent prior to initiation of study procedures
* Patient must be willing to comply with the specified follow-up protocol

Exclusion Criteria:

* In-stent restenotic lesions (ISR occlusions)
* Distal popliteal of 3-vessel tibial occlusion
* Patients on hemodialysis because of heavily calcified vessels
* Recent thrombophlebitis, uremia, or deep venous thrombus (within past 30 days)
* Patients receiving dialysis or immunosuppressant therapy
* Thrombolysis of the target vessel within 72 hours prior to the index procedure with residual intraluminal thrombi
* Recent major stroke within the past 6 months
* Aneurysmal disease of the aorta, iliac, femoral or popliteal arteries
* Required stent placement across or within 0.5 cm of the femoral bifurcation
* Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of a stent device if necessary
* Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, Nitinol (nickel titanium), contrast agent, that cannot be medically managed
* Serum creatinine level >/= 2.5 mg/dl at time of screening visit
* Known or suspected active infection at the time of the procedure
* Bleeding diathesis
* Presence of an aortic, iliac or femoral artificial graft
* Life expectancy less than one year, or any other factors preventing clinical follow-up.
* Use of cryoplasty, laser, or atherectomy devices on the target vessel at the time of index procedure
* Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol
* Patient is known to be pregnant, incarcerated, mentally incompetent, and/or alcohol or drug abuser
* Patient is currently participating in any other investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or future participation in such studies prior to the completion of this study.
* Patient has had major surgical or interventional procedures unrelated to this study within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency | Immediate and at 6 months follow-up
  Primary patency after 6 months follow-up defined as no significant reduction of flow detectable by vascular imaging through the index lesion and without any further clinically driven target vessel revascularization performed in the interim
Primary Patency | 12 months
  Primary patency after 12 months follow-up defined as no significant reduction of flow detectable by vascular imaging through the index lesion and without any further clinically driven target vessel revascularization performed in the interim

SECONDARY OUTCOMES:
Freedom from major adverse event | 30-days to 1year
  30-days, 6 months and 1 year freedom from all causes of death, index limb amputation and target vessel recanalization (TVR)
Binary vessel restenosis | 6 months to 1 year
  6-month and 1-year binary vessel restenosis (>50%) defined by Duplex (≥50% restenosis based on a peak systolic velocity ratio ≥ 2.5), CTA, MRA or DSA according to well-established radiological criteria
Secondary vessel patency | Immediate to 1 year
  Secondary patency up to 12 months follow-up defined as no significant reduction of flow detectable by vascular imaging through the index lesion following the loss of primary patency
AHA Clinical Improvement Score | At 3 months, 6 months and 1 year
QALY estimation | At 6 months and 1 year
  QALY estimation of the two study methods with the use of the SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Siablis, MD, PhD, Principal Investigator — University Hospital of Patras
Locations (5):
- Greece (3):
  - Patras University Hospital, Rio, Achaia
  - Attikon University Hospital, Athens, Attica
  - Heraklion University Hospital, Heraklion
- Insubria University Hospital, Varese, Varese, Italy
- Guy's and St Thomas' Hospitals, NHS Foundation Trust, London, United Kingdom